CLINICAL TRIAL: NCT05651659
Title: Preventing and Approaching Crises for Frail Community-dwelling Patients Through Innovative Care (PRACTIC) - an Effectiveness Study
Brief Title: Preventing and Approaching Crises for Frail Community-dwelling Patients Through Through Innovative Care (PRACTIC)
Acronym: PRACTIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); The Norwegian National Advisory Unit on Ageing and Health (Unknown); Helse Stavanger HF (Other Government); Hochschule für Gesundheit, University of Applied Sciences, Bochum, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 150667
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-03

CONDITIONS: Frailty
Keywords: frailty; crises; home care services; community-dwelling people; behavioural and psychological symptoms of dementia (BPSD); psychosocial interventions; case conferences
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (RCT) with two parallel groups: intervention municipalities and control municipalities
Who Masked: Outcomes Assessor
Masking Description: Specially trained nurses (data assessors) from the project's research centre who are not affiliated with the municipalities will, together with staff members in the home care services, assess patients' baseline characteristics before randomisation. These data assessors will after randomisation be blinded to the randomisation result. They will assess the effect of the intervention via telephone by interviewing the participants, the next of kin and the staff members who know the patient best, at three months and six months after baseline assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventions municipalities (Experimental): Locally adapted TIME (Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms) intervention. Municipalities will be randomly assigned to either the intervention group or the control group. A biostatician will perform the randomisation procedure independently of the project management team and the municipalities. The project management team will provide the home care services in the municipalities with the randomisation and allocation results immediately following this procedure. The intervention will start with the educational sessions (described below) within one to two weeks after randomisation.
  Interventions: Other: TIME model in the prevention and treatment of crises in frail community-dwelling people
- Control municipalities (No Intervention): Care as usual

INTERVENTIONS:
Other: TIME model in the prevention and treatment of crises in frail community-dwelling people — TIME is a manual-based, multicomponent programme that will include a rigorous assessment of the crises, one or more interdisciplinary case conferences and the testing and evaluation of customised treatment measures.This multicomponent interdisciplinary model consisting of three overlapping phases. First the assessment phase where the care staff and the physician collaborate in a comprehensive bio-psychosocial assessment. The second phase is the reflection phase with interdisciplinary case conferences based on principles from cognitive behavioural therapy and abc-method, where a customized treatment plan is developed. The abc-method from cognitive behavioural therapy is used as an analytic tool for the analyses of the complex challenges in the case conferences. In the third phase the treatment plan is implemented and evaluated systematically.
  Arms: Interventions municipalities

SUMMARY:
Preventing and approaching crises for frail community-dwelling patients through innovative care (PRACTIC). Participatory action research in a cluster randomised controlled trial. The primary purpose of this study is to test the effectiveness of an adapted version of a bio-psychosocial person centred model (TIME) to prevent and resolve crises for frail community-dwelling people receiving home care services. The investigators have formulated the following research questions (RQ):

RQ1: Can the TIME model adapted for home care service, prevent, and resolve crises in frail people receiving home care services? RQ2: Which participant characteristics or organizational factors are associated with the effect of the TIME model? RQ3: What are the experiences of the users of home care services on how crises were approached during the trial?

DETAILED DESCRIPTION:
This study is part of the larger PRACTIC (Preventing and approaching crises for frail community-dwelling patients through innovative care) study. This is a six-month cluster randomized controlled trial (RCT). The trial will be conducted in 30 municipalities including 150 frail community-dwelling participants receiving homecare services judged by the services to have imminent crises. The proposed sample of 150 participants is based on a power calculation with clusters of approximately 5 participants from each of the 30 municipalities. Each municipality will be defined as a cluster and will be randomized to receive either the locally adapted TIME intervention (the intervention group) or care as usual (the control group). TIME is a manual-based, multicomponent programme that will include a rigorous assessment of the crises, one or more interdisciplinary case conferences and the testing and evaluation of customised treatment measures. For the interviews in RQ3, the investigators will use a purposeful sample of approximately 15 dyads with 15 patients and next of kin from the intervention municipalities in the RCT

Specially trained nurses (data assessors) from the project's research centre who are not affiliated with the municipalities will, together with staff members in the home care services, assess patients' baseline characteristics before randomisation. The data assessors will assess the effect of the intervention via telephone by interviewing the participants, the next of kin and the staff members who know the patient best, at three months and six months after baseline assessments. The interviews will based on a semi-structured interview guide where the participants will be asked to reflect on two main themes.

To evaluate the effects of a bio-psychosocial intervention like TIME to prevent and resolve crises in a heterogenous population, there is a need for a goal-oriented outcome compromising this variability. The goal of the intervention and the outcome will necessarily vary from patient to patient. The investigators will therefore use a individual goal-oriented interview, the PRACTIC goal-setting interview (PGI), based on The Bangor Goalsetting Interview, BGSI.

ELIGIBILITY:
Inclusion Criteria for patients:

1. in need of home care services
2. a score ≥5 on the Clinical Frailty Scale (indicating mild to severe frailty)
3. perceived by the home care service as being in an unstable situation with a high risk for acute institutionalisation or showing resistance to care.

Exclusion Criteria for patients:

- expected short life expectancy (i.e., <4 weeks).

Inclusion criteria for next of kin (for RQ3):

1. being next of kin of a user of home care services who meets the above mentioned inclusion criteria
2. regular contact with the patient (i.e., at least once a week).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in PGI (PRACTIC Goal-setting Interview) from baseline to 3 months | Change from baseline at 3 months using the PGI (scale of 1-10)
  The primary outcome of the trial is the difference in the change between intervention and control group in individual goal achievement to resolve or reduce the challenges of the crises.

SECONDARY OUTCOMES:
Change in PGI (PRACTIC Goal-setting Interview) | at 6 moths
  the differences in the change between intervention and control group in the BGSI scale at 6 months, in neuropsychiatric symptoms
Change in symptoms (NPS) | at 3 months
  Neuropsychiatric symptoms (NPS) measured by the Neuropsychiatric Inventory (NPI-NH). Score for each symptom: 0-12 points. Total score 144.
Change in symptoms (NPS) | at 6 months
  Neuropsychiatric symptoms (NPS) measured by the Neuropsychiatric Inventory (NPI-NH). Score for each symptom: 0-12 points. Total score 144
Change in quality of life measured | at 3 months
  Quality of life measured by the Quality of Life in Late Stage Dementia scale (QUALID). The score will remain between 11 and 55, with 11 representing the highest quality of life.
Change in quality of life measured | at 6 moths
  Quality of life measured by the Quality of Life in Late Stage Dementia scale (QUALID).The score will remain between 11 and 55, with 11 representing the highest quality of life.
Change in distress perceived by the next of kin | at 3 months
  Distress perceived by the next of kin measured by the Relative Stress Scale (RSS). Total score between 0-60, higher score in an area, more likely higher relative stress.
Change in distress perceived by the next of kin | at 6 months
  Distress perceived by the next of kin measured by the Relative Stress Scale (RSS). Total score between 0-60, higher score in an area, more likely higher relative stress.
Change in rejection of care | at 3 months
  Rejection of care - Minimal Data Set (MDS)
Change in rejection of care | at 6 months
  Rejection of care - Minimal Data Set (MDS)
Change at Activities of Daily Living | at 3 months
  Activities of Daily Living - assessed with the Physical Self-Maintenance Scale (PSMS). Total score between 0-30, higher score in an area, more likely that the patient may be in need of help in that area.
Change at Activities of Daily Living | at 6 months
  Activities of Daily Living - assessed with the Physical Self-Maintenance Scale (PSMS).
  Total score between 0-30, higher score in an area, more likely that the patient may be in need of help in that area.
Change in medication from medical records | at 3 months
  Medication from medical records
Change in medication from medical records | at 6 months
  Medication from medical records
Institutionalization | at 3 months
  Change in level of care
Institutionalization | at 6 months
  Change in level of care
Clinical Frailty scale | 6 months
  Frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
EQ-5D questionnaire | 6 months
  The EQ-5D questionnaire to evaluate pain and discomfort. The dimension pain/discomfort has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement.

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Bergh, MD. PhD, Study Director — Sykehuset Innlandet HF
Locations (1):
- Sykehuset Innlandet, Ottestad, Norway, Norway

IPD SHARING:
Plan to Share IPD: Yes
Collaborating partners in the study will not have access to the individual participant data. The data collected in the study are not publicly available. De-identified participant data will be made available upon reasonable request to the members of the research team at the Research Centre for Age-related Functional Decline and Disease (AFS), Innlandet Hospital Trust.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data and supporting documents are available from 6 December 2024 and will remain available until 1 April 2031.
Access Criteria: De-identified participant data will be made available upon reasonable request from reseachers to the members of the research team at the Research Centre for Age-related Functional Decline and Disease (AFS), Innlandet Hospital Trust.

REFERENCES:
- [Derived] Vaeringstad A, Kirkevold O, Dalbak ETG, Myhre J, Feiring IH, Bergh S, Lichtwarck B. Development of the PRACTIC Goal Setting Interview (PGSI) for Frail Community-Dwelling Patients. Feasibility, Interrater Reliability and Content validity-a Mixed Methods Study. Patient Prefer Adherence. 2025 Dec 12;19:4033-4050. doi: 10.2147/PPA.S557233. eCollection 2025. PMID 41424838
- [Derived] Dalbak ETG, Vaeringstad A, Lichtwarck B, Myhre J, Holle D, Bergh S, Kirkevold O. Preventing and approaching crises for frail community-dwelling patients through innovative care (PRACTIC): study protocol for a process evaluation of a complex intervention in home care service. Trials. 2025 May 28;26(1):178. doi: 10.1186/s13063-025-08876-w. PMID 40437640
- [Derived] Vaeringstad A, Dalbak ETG, Holle D, Myhre J, Kirkevold O, Bergh S, Lichtwarck B. PReventing and Approaching Crises for frail community-dwelling patients Through Innovative Care (PRACTIC): protocol for an effectiveness cluster randomised controlled trial. Trials. 2024 May 6;25(1):304. doi: 10.1186/s13063-024-08117-6. PMID 38711048

DOCUMENTS (1):
  • Study Protocol (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT05651659/Prot_004.pdf